CLINICAL TRIAL: NCT00508508
Title: Mobilizing Peer Support for Effective Heart Failure Self-Management
Brief Title: Effectiveness of Peer Support in Improving Heart Failure Self-Management and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rebecca Mase, Project Manager, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 429; 1R01HL085420-01 (NIH)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; Peer Support; Self Management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Behavioral: IVR
  Interventions: Behavioral: Interactive Voice Response System
- 2 (Experimental): Behavioral: Nurse-Led Group Visits
  Interventions: Behavioral: Nurse-Led Group Clinic Visits

INTERVENTIONS:
Behavioral: Interactive Voice Response System — Participants using IVR will receive training in peer communication techniques and participate in an initial nurse-led interactive group visit. They will then be asked to communicate at least weekly with their partner using the IVR system. The IVR system will also automatically send reminder calls to participants and allow them to leave voice mail messages for their partner and their care manager.
  Other Names: Telephone Peer-Support
  Arms: 1
Behavioral: Nurse-Led Group Clinic Visits — At Months 1, 3, and 6, participants will take part in group visits led by nurses to discuss HF self-management strategies.
  Other Names: Self-Management Group Support and Training
  Arms: 2

SUMMARY:
Heart failure (HF) patients living in low-income or isolated areas may have limited access to necessary clinic services and more difficulty in self-managing their illness. This study will evaluate a program that combines group health care visits and a peer-to-peer telephone buddy system at improving health outcomes among low-income and racial minority HF patients.

DETAILED DESCRIPTION:
HF is a life-threatening condition in which the heart can no longer pump enough blood to the rest of the body. It is important for individuals with heart failure to closely monitor their symptoms, seek out medical attention when appropriate, and effectively self-manage their condition. However, people with HF are often frail, poor, and socially isolated. These factors may limit their ability to access clinic-based services and self-manage their condition. Research has shown that group health care visits with other HF patients and peer support for self-care behaviors are effective at improving heath care outcomes. This study will use an interactive voice response (IVR) system, which is a low-cost telephone system that allows calls to be made through a central 1-800 number, thereby eliminating the need to distribute home phone numbers or pay for long distance calls. Through the IVR system, participants will receive and provide peer support by sharing and discussing HF self-management techniques. The IVR system will also facilitate patient communication with care managers. This study will evaluate the effectiveness of the peer-to-peer IVR program in combination with group health care visits led by HF nurses at reducing hospitalization and death rates among HF patients. Participants will be drawn from a community health care system that primarily serves large numbers of racial minority and socioeconomically vulnerable people.

This study will enroll 288 moderate- to high-risk HF patients from St. Joseph Mercy Health System in Ypsilanti, Michigan. Participants will be paired up with another HF patient, based on gender and illness severity. Each pair will be randomly assigned to receive either usual care or usual care plus the nurse-led group visits and the IVR program. Participants using IVR will receive training in peer communication techniques and participate in an initial nurse-led interactive group visit. They will then be asked to communicate at least weekly with their partner using the IVR system. The IVR system will also automatically send reminder calls to participants and allow them to leave voice mail messages for their partner and their care manager. At Months 1, 3, and 6, participants will take part in group visits led by nurses to discuss HF self-management strategies. Study staff will monitor participants' use of the IVR system, including the dates, duration, and recipients of all phone calls. At Months 6 and 12, all participants will complete questionnaires and undergo a medical record review to assess hospitalization and death rates, quality of life, self-management behaviors, social support, satisfaction with HF care, and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HF
* Inpatient Hospital stay or Heart Failure Clinic Appointment

Exclusion Criteria:

* Serious mental illness or cognitive dysfunction
* Does not speak English fluently
* Receives most HF care outside the St. Joseph Mercy Health System
* Unable to use the telephone to access the IVR system
* Will be discharged to a long-term care or hospice facility
* End-stage cancer or other end-stage condition

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2007-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Re-hospitalization and death rates | Measured at Month 12
Total hospitalizations | Measured at Month 12
HF-specific quality of life | Measured at Months 6 and 12

SECONDARY OUTCOMES:
HF self-management behaviors, treatment regimens, and perceived social support | Measured at Months 6 and 12
HF self-care self-efficacy and autonomous motivation | Measured at Months 6 and 12
Satisfaction with HF care | Measured at Months 6 and 12
Depressive symptoms | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: M.E. Michele Heisler, MD, Principal Investigator — University of Michigan, Ann Arbor, Internal Medicine, General Medicine
Locations (1):
- St. Joseph Mercy Hospital, Ypsilanti, Michigan, United States

REFERENCES:
- [Derived] Heisler M, Halasyamani L, Cowen ME, Davis MD, Resnicow K, Strawderman RL, Choi H, Mase R, Piette JD. Randomized controlled effectiveness trial of reciprocal peer support in heart failure. Circ Heart Fail. 2013 Mar;6(2):246-53. doi: 10.1161/CIRCHEARTFAILURE.112.000147. Epub 2013 Feb 6. PMID 23388114